CLINICAL TRIAL: NCT02190890
Title: Effects of Different Deep Dry Needling Dosages on Pain and Postneedling Soreness in the Treatment of Patients With Cervical Myofascial Pain
Brief Title: Dry Needling Dosage in the Treatment of Myofascial Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16/2013
Record Dates: First submitted 2014-07-04; First posted 2014-07-15 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- Dry needling: 4 local twitch responses (Experimental): Deep dry needling in the active myofascial trigger point in the upper trapezius muscle. The muscle fibers were repeatedly perforated by rapidly inserting and partially withdrawing the needle from the MTrP until 4 local twitch responses were elicited.
  Interventions: Procedure: Dry needling
- Dry needling: 6 local twitch responses (Experimental): Deep dry needling in the active myofascial trigger point in the upper trapezius muscle. The muscle fibers were repeatedly perforated by rapidly inserting and partially withdrawing the needle from the MTrP until 6 local twitch responses were elicited.
  Interventions: Procedure: Dry needling
- Dry needling: Until no more local twitch responses elicited (Experimental): Deep dry needling in the active myofascial trigger point in the upper trapezius muscle. The muscle fibers were repeatedly perforated by rapidly inserting and partially withdrawing the needle from the MTrP until no more local twitch responses were elicited.
  Interventions: Procedure: Dry needling
- Control (Active Comparator): The needle was inserted 1.5 cm away from the trigger point in the trapezius muscle and withdrawn without any consecutive insertion.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Dry needling
  Arms: Dry needling: 4 local twitch responses; Dry needling: 6 local twitch responses; Dry needling: Until no more local twitch responses elicited
Procedure: Control
  Arms: Control

SUMMARY:
The purpose of this study are (1) to determine the effectiveness of different dry needling dosages in the treatment of myofascial trigger points in the upper trapezius muscle in patients with myofascial neck pain, (2) to assess postneedling soreness and tenderness and (3) evaluate the influence of psychological factors on the perception of postneedling soreness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an active myofascial trigger point. Neck pain: Superior to 3 cm in VAS

Exclusion Criteria:

* Neck area: Fracture, radiculopathy, previous surgery, previous needling treatment in the last 6 months, previous analgesic medication (24 hours), psychiatric disease

Ages: 18 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain | 1 week
  Visual analog scale. A 100mm VAS, ranging from 0mm (no pain) to 100mm (worst imaginable pain).
Postneedling soreness | 1 week
  Visual analog scale. A 100mm VAS, ranging from 0mm (no pain) to 100mm (worst imaginable pain).

SECONDARY OUTCOMES:
Pressure pain threshold | 1 week
  Three consecutive trials of pressure pain threshold on the active trigger point at a rate of 1 kg/sec at intervals of 30 seconds were conducted.
Cervical range of motion | 1 week
  The subjects sat in a chair and a CROM goniometer was placed over the head. They were asked to perform active neck movements to the fullest extent of their mobility. Each movement was recorded three times and the average value was calculated.
Neck disability | 1 week
  Neck Disability Index questionnarie was completed.
Pain in cervical range of motion | 1 week
  Pain in a numerical pain rating scale during all cervical movements was recorded.
Psychological factors | Pre-intervention
  State Trait Anxiety Inventory (STAI-T)
Psychological factors | Pre-intervention
  Beck Depression Inventory (BDI-II)
Psychological factors | Pre-intervention
  Tampa Scale for Kinesiophobia
Psychological factors | Pre-intervention
  Pain Catastrophizing Scale

REFERENCES:
- [Derived] Martin-Pintado-Zugasti A, Fernandez-Carnero J, Leon-Hernandez JV, Calvo-Lobo C, Beltran-Alacreu H, Alguacil-Diego I, Gallego-Izquierdo T, Pecos-Martin D. Postneedling Soreness and Tenderness After Different Dosages of Dry Needling of an Active Myofascial Trigger Point in Patients With Neck Pain: A Randomized Controlled Trial. PM R. 2018 Dec;10(12):1311-1320. doi: 10.1016/j.pmrj.2018.05.015. Epub 2018 May 29. PMID 29857165